CLINICAL TRIAL: NCT02913157
Title: Open-label, Single-center, Single-arm Futility Trial Evaluating Oral Hydroxychloroquine 200mg BID for Reducing Progression of Disability in Patients With Primary Progressive Multiple Sclerosis (PPMS)
Brief Title: Hydroxychloroquine in Primary Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Marcus Werner Koch, Assistant Professor, University of Calgary, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCQ_MS01
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis, Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxychloroquine (Experimental): Oral Hydroxychloroquine, 200mg BID
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Orally administered Hydroxychloroquine
  Other Names: Plaquenil

SUMMARY:
The purpose of this clinical trial is to determine if HCQ in a dose of 400mg daily can prevent worsening of walking ability in people PPMS. The number of participants in this study will be 35. A maximum of 42 people with PPMS will be included. The trial is funded through a private donation to the Hotchkiss Brain Institute MS Translational Clinical Trials Research Program and the University of Calgary. There is no sponsorship from the pharmaceutical industry.

DETAILED DESCRIPTION:
In patients with primary progressive multiple sclerosis (PPMS) there is ongoing slow and continuous loss of nerve cells, which causes damage to the brain and spinal cord. This ultimately becomes noticeable as slowly and continuously worsening disability. While the cause of this ongoing damage is unknown, it appears that at least part of the damage may be caused by cells in the brain called "microglia" (a type of immune cell that reside in the brain and spinal cord). These microglial cells can have beneficial roles, for instance when they clear away debris, but they can also cause damage to brain cells. In PPMS, microglial cells are often found to be in a state of activation, and it is currently believed that this constant activation of microglial cells is likely an important cause of the ongoing damage to brain cells.

Current treatments for MS only work in relapsing-remitting MS, and can prevent relapses, but so far there are no treatments that effectively target PPMS. Therapies for PPMS are needed. The investigators believe that treatments that target and reduce the activation of microglial cells may be a useful treatment strategy.

Hydroxychloroquine (HCQ) is a medication that has been shown to decrease the activity of human microglia in laboratory experiments. Animal experiments have also shown that treatment with HCQ can reduce the disease activity of an animal model of MS. HCQ, therefore, may also reduce the activity of microglia in people with PPMS, and hopefully prevent or slow down the progression of disability in PPMS.

HCQ is currently approved in Canada to treat malaria and the rheumatic diseases Systemic Lupus Erythematodes (SLE) and Rheumatoid Arthritis (RA). HCQ is available as a tablet that is usually taken two times per day. Doses up to 600mg per are used in clinical practice, but the investigators estimate that a dose of only 400mg daily, given as two doses of 200mg, will be sufficient to decrease the activity of microglia in patients with PPMS. HCQ is usually well tolerated.

Following a MinMax Simon-2-stage design, the study will require 35 patients with complete 18 month follow-up. Presuming 20% drop-out, the investigators anticipate recruiting up to 42 patients. The trial will be conducted as follows: patients will continuously enter into the study until 35 patients have completed 18 months of follow-up with at least 75% adherence which will be measured by study drug count.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Men and women aged of 18 and 65 years inclusive
* Who are followed at the Calgary MS Clinic
* With Primary Progressive Multiple Sclerosis, according to current diagnostic criteria
* Screening Expanded Disability Status Scale score between 4.0 and 6.5 inclusive.
* Screening timed 25 foot walk (average of two trials) of 5.5 seconds or more.

Exclusion Criteria:

* Patients undergoing treatment with antimalarial drugs, amiodarone, dapsone or digoxin
* Patients with known retinopathy
* Patients whose screening ophthalmological exam shows retinopathy
* Patients whose screening MRI scan shows gadolinium enhancing lesions
* Patients with known renal insufficiency
* Patients with known significant hepatic impairment
* Patients with known porphyria
* Patients with known allergy or other intolerability to HCQ, or to gadolinium MRI contrast agent
* Patients currently using Fampridine or 4-aminopyridine
* Patients planning to start Fampridine or 4-aminopyridine during the study period
* Patients planning to start Baclofen or Tizanidine during the duration of the study
* Patients who increase the dose of Baclofen or Tizanidine during the study period
* Patients who receive treatment with Botulinum toxin in the leg muscles during the study period
* Patients using amiodarone, dapsone, digoxin or antimalarial drugs other than HCQ
* Patients who are unable or unwilling to undergo gadolinium enhanced MRI scans
* Pregnant or breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Timed 25-Foot Walk (T25FW) | Change in Timed 25-Foot Walk performance between the 6 month and 18 month visit.
  quantitative ambulation performance test

SECONDARY OUTCOMES:
9-Hole Peg Test | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  Brief, standardized, quantitative test of upper extremity
Symbol Digit Modalities Test | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  measures cognitive processing speed and working memory
Functional Systems and Expanded Disability Status Scale (EDSS) | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  standard measure of neurologic impairment that is used to describe disability in MS. The neurological assessment comprises seven functional system
Modified Fatigue Impact Scale (MFIS) | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  structured, self-report questionnaire with 21 items concerning how fatigue impact patients quality of life
Multiple Sclerosis Quality of Life Scale 54 item version | baseline, 1 month follow-up, 6 months follow-up, 12 months follow-up, and 18 months follow-up
  54-item multidimensional health-related quality of life measure that combines both generic and MS-specific items

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Koch, Principal Investigator — University of Calgary
Locations (1):
- MS Clinic Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Baeva ME, Tottenham I, Koch M, Camara-Lemarroy C. Biomarkers of disability worsening in inactive primary progressive multiple sclerosis. J Neuroimmunol. 2024 Feb 15;387:578268. doi: 10.1016/j.jneuroim.2023.578268. Epub 2023 Dec 23. PMID 38157653
- [Derived] Camara-Lemarroy C, Silva C, Gohill J, Yong VW, Koch M. Serum neurofilament-light and glial fibrillary acidic protein levels in hydroxychloroquine-treated primary progressive multiple sclerosis. Eur J Neurol. 2023 Jan;30(1):187-194. doi: 10.1111/ene.15588. Epub 2022 Oct 25. PMID 36214614
- [Derived] Brown D, Moezzi D, Dong Y, Koch M, Yong VW. Combination of Hydroxychloroquine and Indapamide Attenuates Neurodegeneration in Models Relevant to Multiple Sclerosis. Neurotherapeutics. 2021 Jan;18(1):387-400. doi: 10.1007/s13311-020-01002-5. Epub 2021 Jan 6. PMID 33410109